CLINICAL TRIAL: NCT02260349
Title: Interest of Indocyanine Green in the Neoplastic Prostatic Tissue Characterization and the Peroperative Surgical Margins Detection During a Radical Prostatectomy.
Brief Title: Interest of Indocyanine Green in Neoplastic Prostatic Tissue
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Scientific coordinator left the hospital
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1308190; 2014-000218-67 (EudraCT Number)
Record Dates: First submitted 2014-09-25; First posted 2014-10-09 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; Prostate cancer; surgical margins; indocyanine green; characterization; prostatectomy; peroperative; detection
MeSH Terms: conditions — Prostatic Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient with Indocyanine green infusion (Experimental): Infusion of Indocyanine Green 0,25 mg/Kg 24h before prostatic surgery
  Interventions: Drug: indocyanine green infusion

INTERVENTIONS:
Drug: indocyanine green infusion — intravenous injection (0,25mg/kg) of the indocyanine green 24h before prostatic surgery.

SUMMARY:
Prostate cancer, with more than 70,000 new cases and 8900 deaths a year in France, is a major public health problem. Until 28% of patients treated with surgery will present a positive surgical margin resulting in an incomplete clearance of the tumoral process and exposing so the patient at a local, systemic recurrence and increased morbidity. An increasing number of international publications have shown (ICG) was interesting for the detection of the sentinel lymph node, in the surgery of tumors of type hepatocarcinoma and liver metastases from colorectal diseases, but also in the surgery of the kidney, bladder or breast. ICG has affinity for tumor and tissues around the tumor related to micro-vascular histology for a localized and specific deposit (EPR effect).

The detection of ICG 's deposits is now possible with to the use of a device which allow to visualize the infra-red fluorescence (NIR; Near Infra-Red) for objects larger than 0.15 mm. Thanks to this feature, the location of residual tumor tissue when performing a radical prostatectomy could be made much easier.

DETAILED DESCRIPTION:
The ability of ICG to detect a surgical margin positive intraoperatively has never be evaluated. We want to perform a monocentric prospective ex-vivo pilot in order to evaluate the diagnostic performance of fluorescence in the detection of surgical margins compared to pathologic analysis. This study will be conducted in 37 patients operated on for a radical prostatectomy after systemic injection of 0, 25 mg/Kg of ICG 24 h before the surgery. The fluorescence analysis will be performed in the operation room and then specimen will be sent to the laboratory for an analysis as usual. Two pieces of prostate will be prelevated according to a protocol. The histopathological procedure will be performed without knowledge of fluorescence analysis. Except the ICG injection the medical procedure won't be changed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostatic cancer proved by biopsy and needing total prostatectomy with or without curettage.
* Patient affiliated to a social security scheme
* Patient has given its informed consent

Exclusion Criteria:

* contra-indication to surgery
* non confirmed adenocarcinoma diagnostic
* antecedent of prostatic cancer treatment
* antecedent of pelvic surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of indocyanine green | 24h after indocyanine green infusion
  Sensitivity (true positive) of the fluorescence due to indocyanine green to detect neoplasm tissue in prostatic biopsy compared to histological analysis

SECONDARY OUTCOMES:
Specificity of indocyanine green | 24h after indocyanine green infusion
  Specificity (true negative) of the fluorescence due to indocyanine green to detect neoplasm tissue in prostatic biopsy compared to histological analysis

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOTTET, PhD, Principal Investigator — CHU SAINT-ETIENNE